CLINICAL TRIAL: NCT06941636
Title: Botulinumtoxin A as a Treatment for Myalgia and Myofacial Pain in Patient With Temporomandibulardisorders - a Quality Study Associated to a New Treatment Routine
Brief Title: Botulinumtoxin A as a Treatment for Myalgia and Myofacial Pain in Patient With Temporomandibulardisorders
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-504033-44-00
Record Dates: First submitted 2024-06-04; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: A randomized doubleblind single-center clinical trial.
Who Masked: Care Provider
Masking Description: The preparation of the drugs and syringe is made by a research assistant.Preparation is performed immediately before the injection. The research assistant will hand over the syringe with the drug to be injected to the investigator to ensure that the patient and the investigator are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BTX-L for myogenous TMD (Active Comparator): Patients (n=45) with myogenious TMD will receive treatment with 50 U of Botox®100 U, AbbVie. The drug will be dissolved in 2 millilitres of room-temperate sterile isotonic saline. This gives 5U/0,1 ml solution and each patient will receive a total o 50 U as described in the protocol
  Interventions: Drug: 5U/0,1 ml Botulinum toxin A
- BTX-H for myogenous TMD (Active Comparator): Patients (n=45) with myogenious TMD will receive treatment with 100 U of Botox®100 U, AbbVie. The drug will be dissolved in 1 millilitre of room-temperate sterile isotonic saline. This gives 10U/0,1 ml solution and each patient will receive a total of 100 U as described in the protocol
  Interventions: Drug: 10U/0,1 ml Botulinum toxin A

INTERVENTIONS:
Drug: 5U/0,1 ml Botulinum toxin A — Botox® 100 U (AbbVie) will be dissolved in 2 milliliters of room-temperature sterile isotonic saline, resulting in a solution concentration of 5 U/0.1 mL. Each patient will receive a total dose of 50 U, administered bilaterally into the masseter and temporalis muscles.
  Other Names: Botox®100 U, AbbVie
  Arms: BTX-L for myogenous TMD
Drug: 10U/0,1 ml Botulinum toxin A — Botox® 100 U (AbbVie) will be dissolved in 1 milliliters of room-temperature sterile isotonic saline, resulting in a solution concentration of 10 U/0.1 mL. Each patient will receive a total dose of 100 U, administered bilaterally into the masseter and temporalis muscles.
  Other Names: Botox®100 U, AbbVie
  Arms: BTX-H for myogenous TMD

SUMMARY:
Both patients and remitters ask for treatment with Botulinumtoxin A (BTX) with the hope that it will be an effective aid for pain, but little is known regarding if the effect is dose dependent.

The aim of this project is to investigate if injections with BTX in the masseter- and temporal muscle is an efficient treatment in patient with myogenous temporomandibular disorders (TMD) and if the effect of BTX is dose dependent.

DETAILED DESCRIPTION:
The primary goal with this study is to expand treatment modalities for patient with myogenous TMD, and to develop clinical protocols with adequate doses for myogenous TMD. A secondary goal is to study if there are differences in treatment effect between sub-groups of myogenous TMD for more personalised pain-treatment.

Hypothesis The investigators hypothesis is that application of BTX into the masseter and temporalis muscle will reduce pain and increase quality of life in patients with myogenous TMD, and that the reduction of pain is only to a certain degree due to the dose. High doses of BTX does not necessarily entail increased reduction of pain or better quality of life. The investigators also hypotheses that the effect may differ in sub-groups of myogenous TMD.

ELIGIBILITY:
Inclusion Criteria:

* Has given a written consent
* Diagnose of myalgia, myofacial pain or myofascial pain with referred pain according
* Average pain due to NRS ≥ 3 for more than three months
* Palpationpain in masseter or temporalis.
* Eventual treatment for orofacial pain > three months ago.
* Adequate contraceptives and a negative pregnancy test.

Patients will still be included even if they have one or more co-diagnoses

* Discdisplacement with or without reduction
* Degenerative joint disease
* Arthralgia

Exclusion Criteria:

* Treatment with BTX during the last 12 months
* Treatment for orofacial pain within the last 3 months.
* Systemic inflammatory diseases (rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis)
* Widespread pain e.g., fibromyalgia
* Neuropathic pain
* Neurologic disease (myasthenia gravis)
* Pain of dental origin
* Use of muscle relaxants, or aminoglycoside antibiotics
* Pregnancy or nursing
* Hypersensitivity to BTX
* Neuropsychiatric conditions.
* Difficulties understanding the Swedish language

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in pain and impact of doses on pain relief | Six months
  Pain level will be assessed using the Numeric rating Scale (NRS, a scale ranging from 0 (no pain) to 10 (worst pain imaginable). A 30% reduction in pain according to the NRS is considered a significant effect. The study compare two doses (low and high)

SECONDARY OUTCOMES:
Changes in quality of life according to The Oral Healthy Impact profile questionnaire (OHIP-5) | 6 months
  The influence of the quality of life will be measured. Scores are categorized as follow: No influence (0-7 p), some influence (8-15 p) and large influence (16-20 p). Higher score mean worse outcomes
Maximum jaw opening in millimeter, with and without pain will be compared to asess treatment outcomes. | 6 months
  Treatment outcome in sub-groups of myogenous TMD.
Changes i pressure pain threshold (PPT) | 6 months
  Sensitivity to pressure induced pain by PPT (pressure pain threshold). PPT will be measured three times and average value will be used.
Changes in psychological factors | 6 months
  According to changes in Axis II (a psykometric form)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica de Flon, Principal Investigator — Region Stockholm
Locations (1):
- Eastman institute Folktandvården Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No